CLINICAL TRIAL: NCT04735718
Title: A Prospective, Open-Label, Pilot, Multicentric Clinical Investigation to Evaluate the Performance and Safety of Cerviron® Ovules in Cervix Lesions Postoperative Care
Brief Title: Clinical Investigation To Evaluate Cerviron Ovules® in Cervix Lesions Postoperative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perfect Care Distribution (Industry)
Collaborators: MDX Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYRON/02/2021
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cervical Lesion
Keywords: cervical lesion

STUDY DESIGN:
Intervention Model Description: A Prospective, Open-Label, Pilot, Multicentric Clinical Investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerviron vaginal ovules (Experimental): Since Cerviron® has an innovative composition, we preferred an exploratory approach for the design of the present clinical investigation. The main objectives and clinical endpoints are the performance and the safety profile of the investigational device.
  Interventions: Device: Cerviron

INTERVENTIONS:
Device: Cerviron — Cerviron® ovules is a class IIb medical device used as adjuvant treatment in cervical lesions of mechanical origin. It favors the healing and re-epithelialization processes and reduces the proliferation of endogenous pathogens.
  Moreover, it provides a strong hemostatic effect, as shown in multiple studies. Moreover, it contains collagen with nutritive, hydrating, healing and trophic effect. Collagen is structurally and functionally a key protein of the extracellular matrix which is also involved in forming the scars during the healing of conjunctive tissues, due to its chemotactic role. Many collagen bandages were developed to improve the repair of the wound, especially of non-infected, chronic, idle cutaneous ulcerations.

SUMMARY:
CYRON is a Prospective, Open-Label, Pilot, Multicentric Clinical Investigation to Evaluate the Performance and Safety of Cerviron® Ovules in Cervix Lesions Postoperative Care. The primary objective is to assess the therapeutic performance and tolerability of Cerviron® Ovules in postoperative care in patients that underwent surgical removal of benign, cervical lesions. The secondary objective of this clinical investigation is the assessment of performance of the medical device by clinical exam and patients' degree of satisfaction related to the use of the medical device.

DETAILED DESCRIPTION:
Identifying premalignant and benign diseases of the cervix and selecting an appropriate treatment path can be challenging. The adult uterine cervix may exhibit a wide variety of pathologic conditions that include benign entities (eg, cervicitis, hyperplasia, nabothian cysts, cervical polyps, leiomyomas, endometriosis, and congenital abnormalities) as well as malignant lesions, particularly cervical carcinoma.

Cervical lesions range from being visible only with an instrument that augments sight such as a colposcope to being visible by speculum examination or endovaginal ultrasound.

The most frequent types of cervical lesions are:

1. Cervical polyp Cervical polyps are benign growths, usually protruding from the surface of the cervical canal. They commonly occur during the reproductive years, especially in women over 20 years of age. Cervical polyps are the most common non-cancerous tumour of the cervix.

The cervical polyps may vary in size, shape, and origin. They can present as single or multiple, tear-shaped or lobular, cherry-red, or greyish-white in color, depending on the vascularity of the lesion. The size of the cervical polyp is typically less than three cm in diameter; however, as mentioned earlier, they can vary in size and can be large enough to fill the vagina or be present at the introitus They usually originate in the endocervical canal. Endocervical polyps may be caused by chronic inflammation. They rarely become malignant.

Nabothian cyst Nabothian cysts are a benign gynecological condition in reproductive age without clinical significance. These cysts are at the squamocolumnar junction of the uterine cervix, which is the targeted anatomical area of brush sampling at the time of cervical screening cytology. They are filled with mucus, but they may also contain proteinaceous material, neutrophils, or neutrophil debris. These cysts usually appear superficially and are easily recognized during colposcopy examination. If left untreated, they can induce considerable enlargement of the cervix, which can lead to symptomatology. Other causes of these large cysts include cystic degeneration of uterine leiomyoma and congenital uterine cysts such as mesonephric and paramesonephric cysts and cystic adenomyosis.

Complications of Nabothian cysts include hematometra, labor passage obstruction, rectal compression, abnormal uterine bleeding, specifically in case of giant cysts, and chronic urinary retention by restricting the bladder's outlet or by compressing the pudendal and sacral nerves, thus, disturbing the nerve supply to the detrusor muscle.

Cervical fibroid Cervical fibroids (myomas) start in the muscle tissue of the cervix. They are similar to uterine fibroids but less common. Cervical fibroids may not cause symptoms. The most common symptom is abnormal vaginal bleeding. Pain during intercourse may happen. If the fibroid becomes large, it may partially block the urinary tract and cause urinary drainage problems such as dribbling or urinary retention. If myomas become infected, they may cause pain, bleeding, or a discharge from the vagina.

The recommended treatment in all cases is excision. After surgery, haemostasis and rapid recovery should be promoted with the support of local, re-epithelizing treatments.

Cerviron® ovules Cerviron® ovules is a class IIb medical device used as adjuvant treatment in cervical lesions of mechanical origin. It favors the healing and re-epithelialization processes and reduces the proliferation of endogenous pathogens.

Bismuth subgallate causes shrinkage of damaged tissue by stopping bleeding and promoting tissue healing. Being an insoluble salt and very little absorbed the bismuth subgalate forms a protective film that allows the other components to act locally. "Through its active ingredient, Bismuth subgallate, Cerviron® ovules exert a protective action on mucous membranes and raw surfaces. Moreover, it provides a strong hemostatic effect, as shown in multiple studies. Moreover, it contains collagen with nutritive, hydrating, healing and trophic effect. Collagen is structurally and functionally a key protein of the extracellular matrix which is also involved in forming the scars during the healing of conjunctive tissues, due to its chemotactic role. Many collagen bandages were developed to improve the repair of the wound, especially of non-infected, chronic, idle cutaneous ulcerations.

The Marigold extract (Calendula Officinalis) contains as active principles carotenoid substances, triterpenic compounds and volatile oil, favouring a healing, antitricomonazic effect and reducing the excessive secretion (leucorrhea). Flavonoids and triterpene glycosides boast soothing properties and also help improve microcirculation. Marigold is mainly used for treating skin disorders: irritation, redness and inflammation. The plant was employed in the civil war to treat wounds.

This is the second clinical investigation on human subjects with this medical device, in which 50 patients will be enlisted, and which will take place in two research centres in Romania.

ELIGIBILITY:
Inclusion Criteria:

* Adult females, aged 18 years to 65 years;
* Subjects presenting benign, ectopic, cervix lesions that were excised no later than 7 days before the Screening Visit, confirmed by colposcopy;
* Subjects presenting a normal cervical cytology report, e.g. Negative for Intraepithelial Lesions or Malignancy (NILM) or slightly modified to Atypical Squamous Cells of Undetermined Significance (ASC-US) in the last 6 months;
* Subjects willing to provide signed informed consent to clinical investigation participation.

Exclusion Criteria:

* Previous history of any malignancy, particularly those that are prone to metastases, including breast, melanoma, gestational trophoblastic disease, and high-grade malignancies of the gastrointestinal tract or lung;
* Subjects with undiagnosed abnormal genital bleeding;
* Subject with vulvar, vaginal or cervical cancer;
* Subjects presenting an abnormal cytology report, e.g. cervical intraepithelial neoplasia" (CIN) or "adenocarcinoma in situ" (AIS) in the last 6 months;
* Watery or foul discharge;
* Subjects with HIV or other immunodeficiency;
* Use of spermicides;
* Use of diaphragm;
* Concomitant topical or systemic anti-infective treatment;
* Unable to comply with visit procedures;
* Subjects included in other clinical investigations with similar objectives

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Clinical Performance Assessed by the Investigator by Colposcopy at End of Treatment Visit | 3 months
  Evolution of cervical lesions at End of Treatment Visit
Rate of treatment-related Adverse Events in subjects participating in the clinical investigation | 3 months
  Number and degree of AE

SECONDARY OUTCOMES:
The Re-epithelialization degree of the cervical mucosa by thorough gynaecological examination (visual evaluation) | at 1, 2 and 3 months
  Gynecological examination by speculum at 1, 2 and 3 months
Evolution of vaginal symptoms and discomfort | at 1, 2 and 3 months
  Presence/absence of symptoms such as pain and/or bleeding at 1, 2 and 3 months
Patient Satisfaction (Likert Scale) | 3 months
  5 point Likert scale to evaluate the degree of satisfaction after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Petrita, CSO, Study Director — MDX Research
Locations (3):
- Romania (3):
  - Institutul National pentru Sanatatea Mamei si Copilului " Alessandrescu-Rusescu", Bucharest
  - Centrul Medical MIȘCĂ, Timișoara
  - Spitalul Clinic Județean de Urgență "Pius Brinzeu", Timișoara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petre I, Toader DO, Petrita R, Pinta AR, Alexa AA, Bita RG. Clinical Performance and Safety of Cerviron(R) Vaginal Ovules in the Management of Symptomatic Cervical Lesions: A National, Multicentric Study. Curr Ther Res Clin Exp. 2024 Oct 9;101:100762. doi: 10.1016/j.curtheres.2024.100762. eCollection 2024. PMID 39717511